CLINICAL TRIAL: NCT01236755
Title: Discontinuation of Orthokeratology on Eyeball Elongation (DOEE) Study. (2) Discontinuation of Lens Wear in New Ortho-k Children
Brief Title: Discontinuation of Lens Wear in New Ortho-k Children (DOEE2)
Acronym: DOEE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Menicon Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-ZG50-2
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Myopia
Keywords: children; corneal reshaping; myopia; myopia progression; orthokeratology
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: All subjects were prescribed with a pair of glasses for seven months and switched to orthokeratology for another seven months
Masking Description: The outcome assessor was responsible for measuring the axial length and was unaware of the intervention (i.e. spectacles or orthokeratology) used by the subjects
Oversight: Data Monitoring Committee: No

ARMS (1):
- ortho-k lenses (Experimental): Children were switched to wear ortho-k lenses for 7 months after wearing single-vision glasses for 7 months
  Interventions: Device: single-vision glasses; Device: ortho-k lenses

INTERVENTIONS:
Device: single-vision glasses — Daily wear of glasses to correct vision in the first seven months of the study
  Other Names: CR-39 lenses
Device: ortho-k lenses — Nightly wear of lenses to correct vision in day time in the second seven months of the study
  Other Names: orthokeratology; corneal reshaping therapy; Menicon Z Night lenses; Menicon Z Night Toric lenses

SUMMARY:
This study aims at investigating the efficacy of myopic control using ortho-k in younger and older children.

DETAILED DESCRIPTION:
Children wearing ortho-k have been shown to have slower rate of myopic progression than those wearing single-vision spectacles (Cho et al. 2005) or soft lenses (Walline et al. 2009). Younger myopic children (aged 6-10 years old) may have the faster increase in myopia than old myopic children (aged 11-15 years old), i.e. the rate of myopic progression may be different in different age groups and in children with different refractive status (Edwards 1999; Fan et al. 2004; Cheng et al. 2007). Although the refractive correction with ortho-k has been well documented, it is unknown whether the efficiency and reversibility of ortho-k for myopic reduction as well as myopic control are similar in children of different age and refractive groups.

In this 14-month study, the eyeball length in 45 younger (6-10 years old) and 45 older (11-15 years old) myopic children before and after ortho-k will be evaluated. Eyeball elongation will be determined for the first 7 months when single-vision glasses will be prescribed (Phase I) and the next 7 months when ortho-k will be prescribed (Phase I). Rate of myopic progression will be determined and compared between the two groups of children in the two phases.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 6 to 15 years old
* Myopia: between 1.50D and 4.50D in at least one eye
* Spherical equivalent (SE): between -1.00D to -4.50D in both eyes
* Astigmatism: ≤ 3.00D of axes 180 +/- 30 or ≤ 1.00D of other axes; and the amount is less than refractive sphere
* Anisometropia: ≤ 1.50D in both refractive sphere, refractive cylinder and SE
* Best corrected monocular visual acuity: equal to or better than 0.10 in logMAR scale in both eyes
* Willingness to wear contact lenses or spectacles on a daily basis
* Can obtain good ortho-k results with the study lenses
* Availability for follow-up for at least 14 months

Exclusion Criteria:

* Strabismus at distance or near
* Contraindication for contact lens wear and ortho-k (e.g. limbus to limbus corneal cylinder and dislocated corneal apex
* Systemic or ocular conditions which may affect contact lens wear (e.g. allergy and medication)
* Systemic or ocular conditions which may affect refractive development (e.g. Down syndrome, ptosis)
* Prior experience with the use of rigid lenses (including ortho-k)
* Prior experience with myopia control treatment (e.g. refractive therapy or progressive spectacles)
* Non-compliance to the follow up schedule
* Non-compliance to the use of the prescribed optical correction
* Poor ocular response to ortho-k lens wear
* Significant residual refractive error after ortho-k treatment resulting in poor unaided vision (worse than 0.18 in logMAR scale)

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Cheng D, Schmid KL, Woo GC. Myopia prevalence in Chinese-Canadian children in an optometric practice. Optom Vis Sci. 2007 Jan;84(1):21-32. doi: 10.1097/01.opx.0000254042.24803.1f. PMID 17220775
- [Background] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Background] Edwards MH. The development of myopia in Hong Kong children between the ages of 7 and 12 years: a five-year longitudinal study. Ophthalmic Physiol Opt. 1999 Jul;19(4):286-94. doi: 10.1046/j.1475-1313.1999.00445.x. PMID 10645384
- [Background] Fan DS, Lam DS, Lam RF, Lau JT, Chong KS, Cheung EY, Lai RY, Chew SJ. Prevalence, incidence, and progression of myopia of school children in Hong Kong. Invest Ophthalmol Vis Sci. 2004 Apr;45(4):1071-5. doi: 10.1167/iovs.03-1151. PMID 15037570
- [Background] Walline JJ, Jones LA, Sinnott LT. Corneal reshaping and myopia progression. Br J Ophthalmol. 2009 Sep;93(9):1181-5. doi: 10.1136/bjo.2008.151365. Epub 2009 May 4. PMID 19416935
- [Result] Cheung SW, Boost MV, Cho P. Pre-treatment observation of axial elongation for evidence-based selection of children in Hong Kong for myopia control. Cont Lens Anterior Eye. 2019 Aug;42(4):392-398. doi: 10.1016/j.clae.2018.10.006. Epub 2018 Oct 24. PMID 30366778

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects in Spectacle and Ortho-k Wearing Phases: Subjects enrolled in the study during the first 7 months in Phase I (daily wear of single-vision spectacles) and the next 7 months in Phase II (nightly wear of orthokeratology lenses)
Period: Spectacles Wearing Phase
Arm/Group | Subjects in Spectacle and Ortho-k Wearing Phases
Started | 91
Completed | 74
Not Completed | 17
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 9
Period: Orthokeratology Wearing Phase
Arm/Group | Subjects in Spectacle and Ortho-k Wearing Phases
Started | 74
Completed | 66
Not Completed | 8
Not completed — Withdrawal by Subject | 5
Not completed — Poor Refractive Correction / Centration | 3

BASELINE CHARACTERISTICS:
Groups:
- Subjects Completed the 14-month Study: Subjects who have completed the study in which they used single-vision spectacles every day for 7 months in Phase I and ortho-k lenses every night for the next 7 months in Phase II to correct their vision.
Arm/Group | Subjects Completed the 14-month Study
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 66

OUTCOME MEASURES:

1. Primary Outcome: Change in Axial Elongation in the Two Study Phases
Description: Axial elongation in children during the two study phases. Phase I: 7 months wearing single-vision spectacles. Phase II: 7 months wearing orthokeratology
Time Frame: 14 months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Axial Elongation in Spectacle and Ortho-k Wearing Phases: Axial elongation in children during the first 7 months in Phase I (daily wear of single-vision spectacles) and the next 7 months in Phase II (nightly wear of orthokeratology lenses)
Arm/Group | Axial Elongation in Spectacle and Ortho-k Wearing Phases
Number analyzed (Participants) | 66
mm
  spectacles wearing phase | 0.163 (0.121)
  orthokeratology wearing phase | 0.047 (0.112)

2. Secondary Outcome: Number of Participants With Serious Adverse Effects
Description: Number of subjects with serious adverse effects of the cornea, the palpebral, bulbar and tarsal conjunctiva
Time Frame: 14 months
Measure: Count of Participants; unit: Participants
Groups:
- Serious Adverse Events in Spectacle and Ortho-k Wearing Phases: Number of subjects with serious adverse events in the cornea and conjunctiva during the first 7 months in Phase I (daily wear of single-vision spectacles) and the next 7 months in Phase II (nightly wear of orthokeratology lenses)
Arm/Group | Serious Adverse Events in Spectacle and Ortho-k Wearing Phases
Number analyzed (Participants) | 66
Participants
  spectacles wearing phase | 0
  orthokeratology wearing phase | 0

ADVERSE EVENTS:
Time Frame: The study started in October 2010 and ended in July 2013. Adverse events during the 33 months were collected and reported
Description: It was a cross-over study in which there was only one Arm/Group. Therefore, the adverse events for the single-vision and orthokeratology phases were combined. The adverse events for each intervention can be found under the second primary outcome in which the results from the two interventions were presented in the two rows
Groups:
- Serious Adverse Events in Spectacle and Ortho-k Wearing Phase: Number of subjects with serious adverse events of the cornea and conjunctiva during the first 7 months in Phase I (daily wear of single-vision spectacles) and the next 7 months in Phase II (nightly wear of orthokeratology lenses)
Arm/Group | Serious Adverse Events in Spectacle and Ortho-k Wearing Phase
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No